CLINICAL TRIAL: NCT05893823
Title: Retrospective Study on Radiological Factors Predictive of Symptomatic Psoas Impingement Development in Protruding Cups in Primary Hip Arthroplasty
Brief Title: Retrospective Study on Radiological Factors Predictive of Psoas Impingement
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: PSOAS IMP
Record Dates: First submitted 2023-05-26; First posted 2023-06-08 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Hip Impingement Syndrome; Prosthetic Complication
Keywords: Iliopsoas Impingement; Overhanging Cup

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients that have symptomatic psoas impingement in a protruding acetabular cup documented by a Pelvis CT scan
  Interventions: Diagnostic Test: Pelvis CT scan
- Controls: Asymptomatic patients with a protruding acetabular cup documented by a Pelvis CT scan
  Interventions: Diagnostic Test: Pelvis CT scan

INTERVENTIONS:
Diagnostic Test: Pelvis CT scan — Post-THA hip pelvis CT scan execution for pain, noise or THA planning for the controlateral hip, with identification of acetabular cup protrusion. Comparation of cases and controls to identify radiological factors that could potentially lead to symptomatic psoas impingement prediction.

SUMMARY:
The purpose of this study is to identify radiological factors on TC of the hip that could lead to prediction of development of symptomatic psoas impingement in patients with protruding acetabular cup after primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip arthroplasty
* Execution of a postoperative Ct scan for pain, noises or planning of the contralateral THA
* 5 years minimum follow-up for the control group, tenotomy of the iliopsoas muscle in the cases group
* Complete clinical and radiological data

Exclusion Criteria:

* Patient's refusal to participate
* Non adequate Ct scans or made for periprosthetic fractures, component mobilization, periprosthetic infection or wearing of the prosthesis
* Incomplete clinical and radiological data
* Inadequate follow-up or regression of the iliopsoas impingement symptoms with non-operative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had undergone a total hip arthroplasty with symptoms of iliopsoas impingement and radiological evidence of a protruding acetabular cup, detected on a Ct scan
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2025-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna
  - IRCCS Istituto Ortopedico Rizzoli, Bologna

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cases | Controls
Started | 35 | 17
Completed | 35 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 35 | 17 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (11.8) | 54.1 (15.3) | 53.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 9 | 29
  Male | 15 | 8 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Cup protrusion [Mean (Standard Deviation); unit: millimeters] — Cup protrusion on sagittal plane and on frontal plane measured in millimeters: from the cup edge to anterior wall, at the center of the head
  millimeters
    Cup protrusion on sagital plane | 12.8 (5.6) | 14.9 (5.4) | 13.5 (5.6)
    Cup protrusion on frontal plane | 5.9 (4.8) | 7.6 (3.4) | 6.4 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Acetabular Cup Antiversion
Description: The angle between the tangent to the cup opening and the tangent to the posterior ischial spines in the axial plane
Time Frame: at baseline (day 0)
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Cases | Controls
Number analyzed (Participants) | 35 | 17
degree | 19.8 (9.5) | 11.5 (9.4)

2. Primary Outcome: Acetabular Cup Inclination
Description: The angle between the tangent to the cup opening and the interteardrop line in the frontal plane
Time Frame: at baseline (day 0)
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Cases | Controls
Number analyzed (Participants) | 35 | 17
degree | 41.8 (6.9) | 43.5 (5.8)

3. Primary Outcome: Femoral Offset
Description: The distance between the center of rotation and the femoral axis in the frontal plane
Time Frame: at baseline (day 0)
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cases | Controls
Number analyzed (Participants) | 35 | 17
millimeters | 40.2 (5.8) | 38.4 (7.7)

4. Primary Outcome: Acetabular Offset
Description: The distance between the center of rotation and the Kohler line in the frontal plane
Time Frame: at baseline (day 0)
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cases | Controls
Number analyzed (Participants) | 35 | 17
millimeters | 32.0 (4.5) | 33.8 (5.6)

5. Primary Outcome: Eccentric Reaming
Description: The distance between the native hip center of rotation and the acetabular cup center of rotation in the axial plane
Time Frame: at baseline (day 0)
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Cases | Controls
Number analyzed (Participants) | 35 | 17
millimeters | 1.8 (4.0) | 0.8 (3.7)

ADVERSE EVENTS:
Time Frame: at baseline (day 0)
Arm/Group | Cases | Controls
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/17
Other Adverse Events (participants affected / at risk) | 0/35 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-14): https://cdn.clinicaltrials.gov/large-docs/23/NCT05893823/Prot_SAP_000.pdf